CLINICAL TRIAL: NCT07245953
Title: A Clinical Study to Evaluate the Efficacy and Safety of HT-101 Injection Combined With HT-102 Injection in Patients With Chronic Hepatitis B
Brief Title: A Clinical Study of HT-101 and HT-102 in Patients With Chronic Hepatitis B Virus Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou HepaThera Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-101&HT-102-201
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (HT-101 + HT-102) (Experimental): Participants will receive HT-101 injection combined with HT-102 injection, administered once every 4 weeks for 24weeks
  Interventions: Drug: HT-101; Drug: HT-102
- Cohort B （placebo；HT-101+HT-102） (Experimental): Participants will receive Placebo injection, administered Q4W for 8 weeks and sequential dosed with HT-101 injection combined with HT-102 injection, administered once every 4 weeks for another 16 weeks
  Interventions: Drug: HT-101; Drug: HT-102; Drug: HT-101 placebo; Drug: HT-102 placebo

INTERVENTIONS:
Drug: HT-101 — HT-101 given by subcutaneous injection
Drug: HT-102 — HT-102 given by subcutaneous injection
Drug: HT-101 placebo — HT-101 placebo given by subcutaneous injection
  Arms: Cohort B （placebo；HT-101+HT-102）
Drug: HT-102 placebo — HT-102 placebo given by subcutaneous injection
  Arms: Cohort B （placebo；HT-101+HT-102）

SUMMARY:
This study is A multicenter, randomized, double-blind, placebo-controlled phase 2 clinical study to evaluate the efficacy and safety of HT-101 injection combined with HT-102 injection in patients with chronic hepatitis B. It consists of two phases: the main trial and the extension period. The main trial phase aims to explore the efficacy of different courses of HT-101 injection combined with HT-102 injection in treating patients with chronic hepatitis B and evaluate the optimal treatment strategy. The extension period phase, based on the main trial, assesses the long-term safety and efficacy of HT-101 injection combined with HT-102 injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were eligible for inclusion into the study if they met each of the following criteria:

Patient with CHB Male subjects weighed ≥ 45.0 kg, female subjects weighed ≥ 40.0 kg, with a body mass index (BMI) between 19.0 and 30.0 kg/m^2 (inclusive); Chronic HBV infection for >/= 6 months; The quantitation level of HBsAg was > 100 IU/mL and <3000 IU/mL; The quantitation level of HBV DNA <LLOQ;

· On Nas therapy for >/= 6 months at the time of screening Subjects promised to use effective contraception for at least 1 month before screening, and have no fertility, donate sperm or eggs and voluntarily take highly effective physical contraception (including partners) during the trial and within 3 months after the end of the trial;

Exclusion Criteria:

* Subjects were excluded from the study if one or more of the following criteria were applicable Participants with history of drug allergy or specific allergy; Participants who had psychiatric conditions or diseases in cardiovascular, respiratory, endocrine, kidney, liver, digestive tract, skin, immune, blood, nerve and other systems; Participants with history of active pathological bleeding, or bleeding tendency; Participants with abnormal results of physical examination, vital sign examination, ECG examination, laboratory test in the screening period which were judged as clinically significant by clinicians; Participants with significant liver fibrosis or cirrhosis; Participants with symptoms or a history of hepatic decompensation; Participants with a history or suspected risk of liver cancer;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving HBsAg < lower limit of detection (LOD) 0.05 International Unit/mL (IU/mL) and HBV DNA < lower limit of quantitation (LLOQ) with or without anti-HBs seroconversion at W60 | From enrollment to the end of treatment at up to 60 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving HBV DNA lower than LLOQ after stopping all anti-HBV treatment | From enrollment to the end of treatment at up to 60 weeks
HBsAg loss rate at W24, W36, W60 | From enrollment to the end of treatment at up to 60 weeks
Maximum Change of Serum HBsAg From Baseline Description | Up to 36 weeks
  Maximum change of serum HBsAg from Day 1 until 36 weeks post last dose (negative values mean reductions from baseline, positive values mean increased from baseline)
Maximum Change of Serum HBV DNA From Baseline Description | Up to 36 weeks.
  Maximum change of serum HBV DNA from Day 1 until 36 weeks (negative values mean reductions from baseline, positive values mean increased from baseline)
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From enrollment to the end of treatment at up to 60 weeks
  Number of subjects with adverse events (AEs) and serious adverse events (SAEs) assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Clinically significant abnormalities | From enrollment to the end of treatment at up to 60 weeks
  Number of subjects with clinically significant abnormalities in vital signs, electrocardiogram (ECG), and laboratory parameters graded by CTCAE v5.0
Maximum Plasma Concentration (Cmax) | HT-101: From predose 1 hour to postdose 8 hours. HT-102: UP to 36 weeks.
  Cmax of HT-101 and its metabolite in plasma. First administration: Predose 1 hour; Postdose 2 hours, 4 hours, 6 hours, 8 hours.
  Changes in the concentration of HT-102 in serum, From Day1 until 36 weeks.
Time to Reach Maximum Plasma Concentration (Tmax) | HT-101: From predose 1 hour to postdose 8 hours. HT-102: UP to 36 weeks.
  Tmax of HT-101 and its metabolite in plasma. First administration: Predose 1 hour; Postdose 2 hours, 4 hours, 6 hours, 8 hours.
  Changes in the concentration of HT-102 in serum, From Day1 until 36 weeks.
Area Under the Plasma Concentration Versus Time Curve (AUC) | HT-101: From predose 1 hour to postdose 8 hours. HT-102: UP to 36 weeks.
  AUC of HT-101 and its metabolite from time 0 to last measurable time. First administration: Predose 1 hour; Postdose 2 hours, 4 hours, 6 hours, 8 hours.
  Changes in the concentration of HT-102 in serum, From Day1 until 36 weeks.
Titers of Anti-drug Antibody (ADA) to HT-102 or HT-101 | UP to 36 weeks
  ADA analysis for predose 36weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, Study Chair — Nanfang Hospital, Southern Medical University
Locations (12):
- China (12):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Ruikang Hospital Affiliated to Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Henan Infectious Diseases Hospital , The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Zhenjiang Third People's Hospital (Zhenjiang Infectious Diseases Hospital), Zhenjiang, Jiangsu
  - Nanchang Ninth Hospital, Nanchang, Jiangxi
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan